CLINICAL TRIAL: NCT02544451
Title: A Phase 3, Rollover Study to Evaluate the Safety and Efficacy of Long-term Treatment With Lumacaftor in Combination With Ivacaftor in Subjects Aged 6 Years and Older With Cystic Fibrosis, Homozygous for the F508del-CFTR Mutation
Brief Title: Rollover Study to Evaluate the Safety and Efficacy of Long-term Treatment With Lumacaftor in Combination With Ivacaftor
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VX15-809-110
Record Dates: First submitted 2015-09-01; First posted 2015-09-09 (Estimated); Results first posted 2019-10-29 (Actual); Last update posted 2021-05-24 (Actual); Status verified 2021-02

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — lumacaftor, ivacaftor drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Treatment Period 1: LUM/IVA to LUM/IVA (Experimental)
  Interventions: Drug: LUM/IVA
- Treatment Period 1: Placebo (PBO) to LUM/IVA (Experimental)
  Interventions: Drug: LUM/IVA
- Treatment Period 1: Observational Cohort (No Intervention)
- Treatment Period 2: LUM/IVA (Experimental)
  Interventions: Drug: LUM/IVA

INTERVENTIONS:
Drug: LUM/IVA — Lumacaftor (LUM) 200 mg every 12 hours (q12h)/ivacaftor (IVA) 250 mg q12h (for 6 through 11 years of age).
  LUM 400 mg q12h/IVA 250 mg q12h (for 12 years and older).
  Other Names: VX-809/VX-770; lumacaftor/ivacaftor
  Arms: Treatment Period 1: LUM/IVA to LUM/IVA; Treatment Period 1: Placebo (PBO) to LUM/IVA
Drug: LUM/IVA — LUM 200 mg q12h/IVA 250 mg q12h (for 6 through 11 years of age).
  Other Names: VX-809/VX-770; lumacaftor/ivacaftor
  Arms: Treatment Period 2: LUM/IVA

SUMMARY:
Study 110 is a Phase 3, multicenter study in subjects aged 6 years and older with cystic fibrosis (CF) who are homozygous for the F508del-CF transmembrane conductance regulator (CFTR) mutation and who participated in Study 109 (NCT02514473) or Study 011B (NCT01897233). Study 110 is designed to evaluate the safety and efficacy of long term treatment of lumacaftor in combination with ivacaftor.

ELIGIBILITY:
Inclusion Criteria:

Subjects entering the Treatment Cohort must meet both of the following criteria:

* Completed study visits up to Week 24 of Study 109 or Week 26 of Study 011B and did not permanently discontinue treatment
* Willing to remain on a stable CF medication through the Safety Follow-up Visit.

Subjects entering the Observational Cohort must meet 1 of the following criteria:

* Completed 24 weeks of study drug treatment in Study 109 or completed 24 weeks of study drug treatment and the Week 26 Safety Follow up in Study 011B.
* Received at least 4 weeks of study drug and completed visits up to Week 24 of Study 109 or Week 26 of Study 011B.

Exclusion Criteria (Treatment Cohort Only):

* History of any comorbidity or laboratory abnormality that, in the opinion of the investigator, might confound the results of the study or pose an additional risk in administering study drug to the subject (e.g., cirrhosis with portal hypertension).
* Pregnant and nursing females.
* Sexually active subjects of reproductive potential who are not willing to follow the contraception requirements.
* History of drug intolerance in the prior study that would pose an additional risk to the subject in the opinion of investigator
* History of poor compliance with study drug and/or procedure in the previous study as deemed by the investigator.
* Participation in an investigational drug trial (including studies investigating lumacaftor and/or ivacaftor).

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 246 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2020-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (60):
- United States (37):
  - Birmingham, Alabama
  - Tucson, Arizona
  - Long Beach, California
  - Palo Alto, California
  - Aurora, Colorado
  - Wilmington, Delaware
  - Jacksonville, Florida
  - Orlando, Florida
  - Atlanta, Georgia
  - Chicago, Illinois
  - Indianapolis, Indiana
  - Iowa City, Iowa
  - Boston, Massachusetts
  - Minneapolis, Minnesota
  - Kansas City, Missouri
  - St Louis, Missouri
  - Omaha, Nebraska
  - Lebanon, New Hampshire
  - Buffalo, New York
  - Syracuse, New York
  - Chapel Hill, North Carolina
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Dayton, Ohio
  - Portland, Oregon
  - Pittsburgh, Pennsylvania
  - Charleston, South Carolina
  - Austin, Texas
  - Houston, Texas
  - Salt Lake City, Utah
  - Colchester, Vermont
  - Charlottesville, Virginia
  - Norfolk, Virginia
  - Richmond, Virginia
  - Seattle, Washington
  - Madison, Wisconsin
  - Milwaukee, Wisconsin
- Australia (5):
  - Parkville, Victoria
  - Herston
  - New Lambton Heights
  - Subiaco
  - Westmead
- Belgium (2):
  - Brussels
  - Leuven
- Canada (3):
  - Vancouver, British Columbia
  - Toronto, Ontario
  - Montreal, Quebec
- Copenhagen, Denmark
- France (3):
  - Bron, Cedex
  - Bordeaux
  - Paris
- Germany (4):
  - Berlin
  - Cologne
  - Giessen
  - Hanover
- Stockholm, Sweden
- United Kingdom (4):
  - Leeds, West Yorkshire
  - Belfast
  - Edinburgh
  - London

REFERENCES:
- [Derived] Chilvers MA, Davies JC, Milla C, Tian S, Han Z, Cornell AG, Owen CA, Ratjen F. Long-term safety and efficacy of lumacaftor-ivacaftor therapy in children aged 6-11 years with cystic fibrosis homozygous for the F508del-CFTR mutation: a phase 3, open-label, extension study. Lancet Respir Med. 2021 Jul;9(7):721-732. doi: 10.1016/S2213-2600(20)30517-8. Epub 2021 Jan 28. PMID 33516285

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study consists of 2 Treatment Periods: Treatment Period 1 and Treatment Period 2. Treatment Period 1 had Treatment Cohorts and an Observational Cohort.
Pre-assignment Details: Participants from Parent Studies 109 (NCT02514473) and 011B (NCT01897233) were enrolled in this study. A total of 240 participants were enrolled in Treatment Period 1 Treatment Cohorts, out of which 1 participant was enrolled but never dosed. Participants enrolled in the Observational and Treatment Period 2 Cohorts were followed for safety endpoint only, no efficacy data were collected.
Groups:
- Treatment Period 1: LUM/IVA to LUM/IVA: Participants received LUM/IVA in parent studies (109, 011B) and continued to receive LUM/IVA for 96 weeks in the current study.
- Treatment Period 1: PBO to LUM/IVA: Participants received placebo (PBO) in parent study (109) and then received LUM/IVA for 96 weeks in the current study.
- Treatment Period 1: Observational Cohort: Participants completed a parent study (109, 011B) but were not eligible or elected to not receive LUM/IVA for 96 weeks in the current study.
- Treatment Period 2: LUM/IVA: Eligible subjects from Treatment Period 1 received LUM/IVA for up to approximately 168 weeks.
Period: Treatment Period 1 (96 Weeks)
Arm/Group | Treatment Period 1: LUM/IVA to LUM/IVA | Treatment Period 1: PBO to LUM/IVA | Treatment Period 1: Observational Cohort | Treatment Period 2: LUM/IVA
Started | 143 | 96 | 6 | 0
Completed | 129 | 84 | 5 | 0
Not Completed | 14 | 12 | 1 | 0
Not completed — Adverse Event | 1 | 6 | 0 | 0
Not completed — Withdrawal of consent (not due to AE) | 3 | 2 | 1 | 0
Not completed — Lost to Follow-up | 2 | 0 | 0 | 0
Not completed — Physician Decision | 4 | 0 | 0 | 0
Not completed — Other | 4 | 4 | 0 | 0
Period: Treatment Period 2 (168 Weeks)
Arm/Group | Treatment Period 1: LUM/IVA to LUM/IVA | Treatment Period 1: PBO to LUM/IVA | Treatment Period 1: Observational Cohort | Treatment Period 2: LUM/IVA
Started | 0 | 0 | 0 | 10
Completed | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 10
Not completed — Commercial drug is available for subject | 0 | 0 | 0 | 10

BASELINE CHARACTERISTICS:
Population: Treatment Cohort: All participants dosed in the parent studies and dosed in the current study.
  Observational Cohort: All participants enrolled in the observational cohort of the current study.
Groups:
- LUM/IVA to LUM/IVA: Participants received LUM/IVA in parent studies (109, 011B) and continued to receive LUM/IVA for 96 weeks in the current study.
- PBO to LUM/IVA: Participants received PBO in parent study (109) and then received LUM/IVA for 96 weeks in the current study.
- Observational Cohort: Participants completed a parent study (109, 011B) but were not eligible or elected to not receive LUM/IVA for 96 weeks in the current study.
- Total: Total of all reporting groups
Arm/Group | LUM/IVA to LUM/IVA | PBO to LUM/IVA | Observational Cohort | Total
Number analyzed (Participants) | 143 | 96 | 6 | 245
Age, Customized [Count of Participants; unit: Participants]
  Less than 9 Years | 58 | 38 | 5 | 101
  Greater than or equal to 9 years | 85 | 58 | 1 | 144
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 83 | 56 | 2 | 141
  Male | 60 | 40 | 4 | 104
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 0 | 4
  Not Hispanic or Latino | 139 | 93 | 6 | 238
  Unknown or Not Reported | 2 | 1 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 140 | 92 | 6 | 238
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 3 | 3 | 0 | 6

OUTCOME MEASURES:

1. Primary Outcome: Treatment Period 1 (Treatment Cohorts): Safety and Tolerability as Assessed by Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Time Frame: Day 1 up to Week 100
Population: Safety set included all participants who received at least 1 dose of study drug in Treatment Period 1.
Measure: Number; unit: participants
Arm/Group | LUM/IVA to LUM/IVA | PBO to LUM/IVA
Number analyzed (Participants) | 143 | 96
participants
  Participants with any AEs | 142 | 94
  Participants with SAEs | 43 | 29

2. Secondary Outcome: Absolute Change in Lung Clearance Index (LCI) 2.5
Description: LCI 2.5 represents the number of lung turnovers required to reduce the end tidal inert gas concentration to 1/40th of its starting value.
Time Frame: From Parent Study Baseline at Week 96
Population: LCI set includes all participants enrolled and dosed in either parent study 109 or 011B LCI sub-study. Analysis period includes both parent study and current study.
Measure: Least Squares Mean (95% Confidence Interval); unit: lung clearance index
Groups:
- LUM/IVA to LUM/IVA: All participants in the LCI set who received LUM/IVA in the parent study.
- PBO to LUM/IVA: All participants in the LCI set who received PBO in the parent study.
Arm/Group | LUM/IVA to LUM/IVA | PBO to LUM/IVA
Number analyzed (Participants) | 133 | 101
lung clearance index | -0.85 [-1.25 to -0.45] | -0.86 [-1.33 to -0.38]

3. Secondary Outcome: Absolute Change in Sweat Chloride
Description: Sweat samples were collected using an approved collection device.
Time Frame: From Parent Study Baseline at Week 96
Population: Full Analysis Set (FAS) includes all participants enrolled and dosed in either parent study. Analysis period includes both parent study and current study.
Measure: Least Squares Mean (95% Confidence Interval); unit: millimole per liter (mmol/L)
Groups:
- LUM/IVA to LUM/IVA: All participants in the FAS who received LUM/IVA in the parent study.
- PBO to LUM/IVA: All participants in the FAS who received PBO in the parent study.
Arm/Group | LUM/IVA to LUM/IVA | PBO to LUM/IVA
Number analyzed (Participants) | 161 | 101
millimole per liter (mmol/L) | -22.9 [-25.5 to -20.3] | -22.8 [-26.3 to -19.3]

4. Secondary Outcome: Absolute Change in Body Mass Index (BMI)
Description: BMI was defined as weight in kilograms divided by height in square meter (m^2).
Time Frame: From Parent Study Baseline at Week 96
Population: FAS.
Measure: Least Squares Mean (95% Confidence Interval); unit: kg/m^2
Arm/Group | LUM/IVA to LUM/IVA | PBO to LUM/IVA
Number analyzed (Participants) | 161 | 101
kg/m^2 | 1.78 [1.56 to 1.99] | 2.04 [1.77 to 2.31]

5. Secondary Outcome: Absolute Change in Cystic Fibrosis Questionnaire-Revised (CFQ-R) Respiratory Domain Score
Description: The CFQ-R is a validated participant-reported outcome measuring health-related quality of life for participants with cystic fibrosis. Respiratory domain assessed respiratory symptoms, score range: 0-100; higher scores indicating fewer symptoms and better health-related quality of life.
Time Frame: From Parent Study Baseline at Week 96
Population: FAS.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | LUM/IVA to LUM/IVA | PBO to LUM/IVA
Number analyzed (Participants) | 161 | 101
units on a scale | 7.4 [4.8 to 10.0] | 6.6 [3.1 to 10.0]

6. Secondary Outcome: Observational Cohort: Safety as Assessed by Serious Adverse Events (SAEs)
Time Frame: Day 1 up to Week 100
Population: All participants included in the observational cohort.
Measure: Number; unit: participants
Arm/Group | Observational Cohort
Number analyzed (Participants) | 6
participants | 1

7. Secondary Outcome: Absolute Change in LCI 5.0
Description: LCI 5.0 represents the number of lung turnovers required to reduce the end tidal inert gas concentration to 1/20th of its starting value.
Time Frame: From Parent Study Baseline at Week 96
Population: LCI set.
Measure: Least Squares Mean (95% Confidence Interval); unit: lung clearance index
Arm/Group | LUM/IVA to LUM/IVA | PBO to LUM/IVA
Number analyzed (Participants) | 133 | 101
lung clearance index | -0.21 [-0.36 to -0.06] | -0.31 [-0.49 to -0.13]

8. Secondary Outcome: Absolute Change in Percent Predicted Forced Expiratory Volume in 1 Second (ppFEV1)
Description: FEV1 is the volume of air that can forcibly be blown out in one second, after full inspiration.
Time Frame: From Parent Study Baseline at Week 96
Population: FAS.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent predicted of FEV1
Arm/Group | LUM/IVA to LUM/IVA | PBO to LUM/IVA
Number analyzed (Participants) | 161 | 101
percent predicted of FEV1 | 3.1 [1.0 to 5.1] | 0.0 [-2.7 to 2.7]

9. Secondary Outcome: Relative Change in ppFEV1
Description: FEV1 is the volume of air that can forcibly be blown out in one second, after full inspiration.
Time Frame: From Parent Study Baseline at Week 96
Population: FAS.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | LUM/IVA to LUM/IVA | PBO to LUM/IVA
Number analyzed (Participants) | 161 | 101
percent change | 4.9 [2.2 to 7.5] | 0.5 [-2.9 to 4.0]

10. Secondary Outcome: Absolute Change in BMI-for-age Z-score
Description: BMI was defined as weight in kilograms divided by height in m^2. z-score is a statistical measure to describe whether a mean was above or below the standard. A z-score of 0 is equal to the mean and is considered normal. Lower numbers indicate values lower than the mean and higher numbers indicate values higher than the mean.
Time Frame: From Parent Study Baseline at Week 96
Population: FAS.
Measure: Least Squares Mean (95% Confidence Interval); unit: z-score
Arm/Group | LUM/IVA to LUM/IVA | PBO to LUM/IVA
Number analyzed (Participants) | 161 | 101
z-score | 0.17 [0.08 to 0.26] | 0.31 [0.19 to 0.42]

11. Secondary Outcome: Absolute Change in Weight
Time Frame: From Parent Study Baseline at Week 96
Population: FAS.
Measure: Least Squares Mean (95% Confidence Interval); unit: kg
Arm/Group | LUM/IVA to LUM/IVA | PBO to LUM/IVA
Number analyzed (Participants) | 161 | 101
kg | 10.3 [9.6 to 11.0] | 11.0 [10.1 to 11.8]

12. Secondary Outcome: Absolute Change in Weight-for-age Z-score
Description: z-score is a statistical measure to describe whether a mean was above or below the standard. A z-score of 0 is equal to the mean and is considered normal. Lower numbers indicate values lower than the mean and higher numbers indicate values higher than the mean.
Time Frame: From Parent Study Baseline at Week 96
Population: FAS.
Measure: Least Squares Mean (95% Confidence Interval); unit: z-score
Arm/Group | LUM/IVA to LUM/IVA | PBO to LUM/IVA
Number analyzed (Participants) | 161 | 101
z-score | 0.12 [0.04 to 0.20] | 0.24 [0.14 to 0.34]

13. Secondary Outcome: Absolute Change in Height
Time Frame: From Parent Study Baseline at Week 96
Population: FAS.
Measure: Least Squares Mean (95% Confidence Interval); unit: centimeter (cm)
Arm/Group | LUM/IVA to LUM/IVA | PBO to LUM/IVA
Number analyzed (Participants) | 161 | 101
centimeter (cm) | 13.4 [12.9 to 14.0] | 13.5 [12.8 to 14.1]

14. Secondary Outcome: Absolute Change in Height-for-age Z-score
Description: as for outcome 12
Time Frame: From Parent Study Baseline at Week 96
Population: FAS.
Measure: Least Squares Mean (95% Confidence Interval); unit: z-score
Arm/Group | LUM/IVA to LUM/IVA | PBO to LUM/IVA
Number analyzed (Participants) | 161 | 101
z-score | -0.01 [-0.08 to 0.07] | 0.02 [-0.07 to 0.11]

15. Secondary Outcome: Absolute Change in Treatment Satisfaction Questionnaire for Medication (TSQM) Total Domain Score
Description: The TSQM measures participants' experiences with their medication on four dimensions: effectiveness, side effects, convenience and global satisfaction. For each dimension, responses are added and transformed in the total domain score, which ranges from 0 to 100, where higher scores indicate greater satisfaction.
Time Frame: From Parent Study Baseline at Week 96
Population: FAS.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | LUM/IVA to LUM/IVA | PBO to LUM/IVA
Number analyzed (Participants) | 161 | 101
units on a scale | 5.1 [1.7 to 8.4] | 3.9 [-0.6 to 8.5]

16. Secondary Outcome: Time-to-first Pulmonary Exacerbation
Description: Pulmonary exacerbation was defined as the treatment with new or changed antibiotic therapy (intravenous, inhaled, or oral) for greater than or equal to 4 sinopulmonary signs/symptoms.
Time Frame: From Parent Study Baseline through Week 96
Population: Analysis included all participants dosed in parent study 109. LUM/IVA to LUM/IVA analysis period includes both parent study and current study. PBO to LUM/IVA analysis period includes the current study only.
Measure: Median (Inter-Quartile Range); unit: days
Groups:
- LUM/IVA to LUM/IVA: All participants who received LUM/IVA in parent study 109.
- PBO to LUM/IVA: All participants who received PBO in parent study 109.
Arm/Group | LUM/IVA to LUM/IVA | PBO to LUM/IVA
Number analyzed (Participants) | 103 | 96
days | 720.00 [278.00 to NA] — Upper limit of inter-quartile range could not be estimated because less than 75% of participants had events. | NA [513.00 to NA] — Median and upper limit of inter-quartile range could not be estimated because less than 50% of participants had events.

17. Secondary Outcome: Percentage of Participants Having At Least 1 Pulmonary Exacerbation Event
Description: as for outcome 16
Time Frame: From Parent Study Baseline through Week 96
Population: as for outcome 16
Measure: Number; unit: percentage of participants
Arm/Group | LUM/IVA to LUM/IVA | PBO to LUM/IVA
Number analyzed (Participants) | 103 | 96
percentage of participants | 49.5 | 32.3

18. Secondary Outcome: Number of Pulmonary Exacerbation Events Per Patient-year
Description: as for outcome 16
Time Frame: From Parent Study Baseline through Week 96
Population: as for outcome 16
Measure: Number (95% Confidence Interval); unit: events per patient-year
Arm/Group | LUM/IVA to LUM/IVA | PBO to LUM/IVA
Number analyzed (Participants) | 103 | 96
events per patient-year | 0.45 [0.33 to 0.61] | 0.30 [0.21 to 0.43]

19. Secondary Outcome: Rate of Change in LCI 2.5
Description: Rate of change analysis evaluates the change in LCI 2.5 after long term treatment with LUM/IVA. A rate of change equal to zero would indicate that treatment effects were stable.
Time Frame: Day 15 after first dose of LUM/IVA through Week 96
Population: As pre-specified in the SAP, this analysis was conducted in the LUM/IVA Overall group because of sample size. Analysis period is 15 days after first dose of LUM/IVA in parent study or current study (if assigned to placebo in study 109) through the end of current study.
Measure: Number (95% Confidence Interval); unit: slope
Groups:
- LUM/IVA Overall: All participants who received LUM/IVA in parent study 109, 011B LCI sub-study, or current study.
Arm/Group | LUM/IVA Overall
Number analyzed (Participants) | 229
slope | -0.01 [-0.12 to 0.09]

20. Secondary Outcome: Rate of Change in LCI 5.0
Description: Rate of change analysis evaluates the change in LCI 5.0 after long term treatment with LUM/IVA. A rate of change equal to zero would indicate that treatment effects were stable.
Time Frame: Day 15 after first dose of LUM/IVA through Week 96
Population: as for outcome 19
Measure: Number (95% Confidence Interval); unit: slope
Arm/Group | LUM/IVA Overall
Number analyzed (Participants) | 229
slope | 0.00 [-0.04 to 0.04]

21. Secondary Outcome: Rate of Change in ppFEV1
Description: Rate of change analysis evaluates the change in ppFEV1 after long term treatment with LUM/IVA. A rate of change equal to zero would indicate that treatment effects were stable.
Time Frame: Day 15 after first dose of LUM/IVA through Week 96
Population: as for outcome 19
Measure: Number (95% Confidence Interval); unit: slope
Groups:
- LUM/IVA Overall: All participants who received LUM/IVA in either parent study or current study.
Arm/Group | LUM/IVA Overall
Number analyzed (Participants) | 257
slope | 0.58 [0.02 to 1.14]

22. Secondary Outcome: Treatment Period 2: Safety and Tolerability as Assessed by Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Time Frame: Day 1 up to Week 168
Population: Safety set included all participants who received at least 1 dose of study drug in Treatment Period 2.
Measure: Number; unit: participants
Arm/Group | Treatment Period 2: LUM/IVA
Number analyzed (Participants) | 10
participants
  Participants with any AEs | 9
  Participants with SAEs | 0

ADVERSE EVENTS:
Time Frame: Treatment Period 1: Day 1 up to Week 100, Treatment Period 2: Day 1 up to Week 168
Description: Only serious adverse events were collected for the observational cohort. Non-serious AEs were not collected and are not reported for the observational cohort. Adverse events reported based on MedDRA version 21.0 for Treatment Period 1 and MedDRA version 22.1 for Treatment Period 2.
Groups:
- Treatment Period 1: PBO to LUM/IVA: Participants received PBO in parent study (109) and then received LUM/IVA for 96 weeks in the current study.
Arm/Group | Treatment Period 1: LUM/IVA to LUM/IVA | Treatment Period 1: PBO to LUM/IVA | Treatment Period 1: Observational Cohort | Treatment Period 2: LUM/IVA
All-Cause Mortality (participants affected / at risk) | 0/143 | 0/96 | 0/6 | 0/10
Serious Adverse Events (participants affected / at risk) | 43/143 | 29/96 | 1/6 | 0/10
Other Adverse Events (participants affected / at risk) | 141/143 | 93/96 | 0/0 | 9/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Period 1: LUM/IVA to LUM/IVA (N=143) | Treatment Period 1: PBO to LUM/IVA (N=96) | Treatment Period 1: Observational Cohort (N=6) | Treatment Period 2: LUM/IVA (N=10)
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 34 | 15 | 1 | 0
Bronchopulmonary aspergillosis allergic (Infections and infestations) | 2 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 1 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 1 | 0 | 0
Atypical mycobacterial lower respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 0 | 0
Lower respiratory tract infection bacterial (Infections and infestations) | 1 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Pulmonary function test decreased (Investigations) | 2 | 2 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 2 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 2 | 0 | 0
Pseudomonas test positive (Investigations) | 1 | 1 | 0 | 0
Atypical mycobacterium test positive (Investigations) | 1 | 0 | 0 | 0
Oxygen saturation decreased (Investigations) | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 4 | 0 | 0 | 0
Distal intestinal obstruction syndrome (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Cystic fibrosis hepatic disease (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0
Cystic fibrosis lung (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 0
Intentional overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Lymphadenitis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Autoimmune hepatitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Period 1: LUM/IVA to LUM/IVA (N=143) | Treatment Period 1: PBO to LUM/IVA (N=96) | Treatment Period 1: Observational Cohort (N=0) | Treatment Period 2: LUM/IVA (N=10)
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 59 | 34 | NA | 4
Upper respiratory tract infection (Infections and infestations) | 36 | 13 | NA | 0
Nasopharyngitis (Infections and infestations) | 21 | 16 | NA | 3
Viral upper respiratory tract infection (Infections and infestations) | 21 | 14 | NA | 0
Sinusitis (Infections and infestations) | 17 | 8 | NA | 0
Otitis media (Infections and infestations) | 13 | 8 | NA | 0
Pharyngitis streptococcal (Infections and infestations) | 12 | 6 | NA | 0
Bacterial disease carrier (Infections and infestations) | 11 | 6 | NA | 2
Influenza (Infections and infestations) | 11 | 6 | NA | 0
Ear infection (Infections and infestations) | 9 | 7 | NA | 1
Rhinitis (Infections and infestations) | 9 | 7 | NA | 6
Upper respiratory tract infection bacterial (Infections and infestations) | 8 | 1 | NA | 0
Bronchitis (Infections and infestations) | 7 | 7 | NA | 2
Pharyngitis (Infections and infestations) | 5 | 7 | NA | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 91 | 64 | NA | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 34 | 21 | NA | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 32 | 18 | NA | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 24 | 13 | NA | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 19 | 15 | NA | 0
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 18 | 7 | NA | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 12 | 4 | NA | 0
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 9 | 3 | NA | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 8 | 1 | NA | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 8 | 4 | NA | 1
Respiration abnormal (Respiratory, thoracic and mediastinal disorders) | 7 | 7 | NA | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 5 | 5 | NA | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 6 | NA | 0
Vomiting (Gastrointestinal disorders) | 30 | 15 | NA | 0
Abdominal pain upper (Gastrointestinal disorders) | 22 | 20 | NA | 0
Abdominal pain (Gastrointestinal disorders) | 17 | 19 | NA | 1
Diarrhoea (Gastrointestinal disorders) | 16 | 8 | NA | 1
Nausea (Gastrointestinal disorders) | 13 | 11 | NA | 1
Constipation (Gastrointestinal disorders) | 11 | 11 | NA | 1
Flatulence (Gastrointestinal disorders) | 4 | 6 | NA | 0
Bacterial test positive (Investigations) | 30 | 16 | NA | 0
Alanine aminotransferase increased (Investigations) | 22 | 21 | NA | 0
Aspartate aminotransferase increased (Investigations) | 17 | 13 | NA | 0
Pseudomonas test positive (Investigations) | 10 | 3 | NA | 0
Pulmonary function test decreased (Investigations) | 8 | 11 | NA | 0
Activated partial thromboplastin time prolonged (Investigations) | 6 | 6 | NA | 0
Forced expiratory volume decreased (Investigations) | 6 | 13 | NA | 1
International normalised ratio increased (Investigations) | 4 | 6 | NA | 0
Prothrombin time prolonged (Investigations) | 3 | 6 | NA | 0
Weight decreased (Investigations) | 1 | 5 | NA | 1
Pyrexia (General disorders) | 45 | 27 | NA | 1
Fatigue (General disorders) | 10 | 11 | NA | 0
Chest pain (General disorders) | 2 | 5 | NA | 0
Headache (Nervous system disorders) | 29 | 26 | NA | 1
Dizziness (Nervous system disorders) | 6 | 5 | NA | 0
Ear pain (Ear and labyrinth disorders) | 12 | 4 | NA | 0
Rash (Skin and subcutaneous tissue disorders) | 10 | 10 | NA | 0
Seasonal allergy (Immune system disorders) | 8 | 5 | NA | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 5 | NA | 1
Decreased appetite (Metabolism and nutrition disorders) | 3 | 6 | NA | 0
Ligament sprain (Injury, poisoning and procedural complications) | 4 | 2 | NA | 1
Pulmonary imaging procedure abnormal (Investigations) | 0 | 0 | NA | 1
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | NA | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 | 2 | NA | 2
Lower respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | NA | 1
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | NA | 1
Rales (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | NA | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 4 | 4 | NA | 1
Eyelid oedema (Eye disorders) | 0 | 0 | NA | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | NA | 1
Gastritis (Gastrointestinal disorders) | 0 | 1 | NA | 1
Hepatomegaly (Hepatobiliary disorders) | 1 | 0 | NA | 1
Glucose tolerance impaired (Metabolism and nutrition disorders) | 1 | 1 | NA | 1
Gastroenteritis (Infections and infestations) | 7 | 4 | NA | 1
Oral fungal infection (Infections and infestations) | 2 | 0 | NA | 1
Respiratory tract infection bacterial (Infections and infestations) | 3 | 1 | NA | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2015-09-15): https://cdn.clinicaltrials.gov/large-docs/51/NCT02544451/Prot_000.pdf
  • Statistical Analysis Plan (2018-07-20): https://cdn.clinicaltrials.gov/large-docs/51/NCT02544451/SAP_001.pdf